CLINICAL TRIAL: NCT00548613
Title: Phase I Study to Determine the Safety and Feasibility of the Use of a Combination Stem Cell Therapy in Patients With Acute Myocardial Infarction
Brief Title: Combination Stem Cell (MESENDO) Therapy for Utilization and Rescue of Infarcted Myocardium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TCA Cellular Therapy (Industry)
Responsible Party: Gabriel P. Lasala, MD, TCA Cellular Therapy, LLC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-02-I
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Coronary Artery Disease; Coronary Arteriosclerosis; Coronary Atherosclerosis; Coronary Disease
Keywords: Myocardial Infarction; Heart Attack; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients with documented acute myocardial infarction (heart attack) occurring within 4-24 hours after onset of symptoms
  Interventions: Biological: MESENDO
- B (Experimental): Candidates for coronary artery bypass grafting that suffered a myocardial infarction (heart attack) within the past 12 months
  Interventions: Biological: MESENDO

INTERVENTIONS:
Biological: MESENDO — Intracoronary transplantation of autologous stem cells via balloon catheter
  Arms: A
Biological: MESENDO — Intracardiac transplantation of autologous stem cells via direct injection
  Arms: B

SUMMARY:
The purpose of this research study is to determine if the transplant of a combination of stem cells, obtained from the bone marrow of the same patient, is effective for utilization and rescue of infarcted myocardium. End points will be the assessment of development of mature and stable new blood vessels as well as improvement in cardiac function.

This, Phase I, single center, prospective, non-randomized, open-label study will evaluate the safety and feasibility of use of the proposed combination of autologous stem cells. Potential subjects who fulfill clinical and laboratory entry criteria at screening will undergo a process of bone marrow aspiration for preparation of the two types of bone marrow-derived stem /progenitor cells to use. The two bone marrow-derived cell types will be mixed and implanted to patients approximately 2 weeks after bone marrow aspiration. After transplant, patients will be have a 3 month follow-up to evaluate safety as well as functional heart improvement by analysis of symptoms, myocardial perfusion SPECT, and echocardiography.

Study population will include adult male and female subjects, ages 18-70, presenting with acute myocardial infarction and subjects who have had a recent (within 12 months) myocardial infarction and will undergo coronary artery bypass grafting.

Patients will be divided in two groups:

* the first group will enroll patients with acute myocardial infarction whom percutaneous coronary intervention restored myocardial flow after 4 hours or greater of the initiation of symptoms,
* the second group will enroll patients who are candidates for coronary artery bypass surgery and had a myocardial infarction in the past 12 months.

Patients will receive the cell mixture by intracoronary or intramyocardial infusion, respectively.

The rationale of this clinical study is based on the observation that most attempts using adult stem cells for myocardial regeneration have utilized a source of bone marrow derived progenitor cells with the potential to generate new blood vessel and thus contribute to the revascularization of the ischemic tissue. This therapy seems to be adequate but not sufficient, since it lacks a source of stem cells capable of differentiating and maturing into cardiac muscle cells, thus contributing to the recovery of local contractility. The proposed combination stem/progenitor cell therapy to be used in this protocol is aimed at contributing cell types capable of regenerating both blood vessels and muscle tissues damaged after MI.

ELIGIBILITY:
Inclusion Criteria:

ARM: A -

* Patients with acute myocardial infarction with ST elevation who underwent percutaneous revascularization between 4 and 24 hours after the initiation of symptoms.

  1. Able to give written informed consent
  2. Age: 18 to 70 years
  3. Gender: Male and Female
  4. Acute myocardial infarction occurring within 4-24 hours after onset of symptoms documented by at least one of the following:

     1. ST Segment elevation greater than 2mm in two or more consecutive leads
     2. New Bundle Branch Block with symptoms consistent of MI
     3. Troponin I greater than 2.0 ng/ml (Normal Range 0 - 1.5 ng/ml)
     4. Totally occluded artery as visualized by angiography

ARM - B

Patients who are candidates for coronary artery bypass grafting surgery according to ACC/AHA guidelines and have had a myocardial infarction in the past 12 months.

1. Able to give written informed consent
2. Patients with coronary artery disease who need coronary artery bypass surgery according to ACC/AHA guidelines
3. Patients with Left Ventricular Ejection Fraction £ 40%.
4. NYHA symptoms Class II (dyspnea with moderate effort)
5. Defined region of myocardial dysfunction related to previous myocardial infarction (within the past 12 months) involving the anterior, lateral, posterior or inferior walls by either of the followings: echocardiography, ventriculography, MRI, or SPECT.
6. Age: 18 to 70 years
7. Gender: Male and Female

Exclusion Criteria:

ARM - A

1. Pregnancy
2. Previous angiogenic therapy or myocardial laser therapy
3. History of cancer within 5 years
4. Known sensitivity to gentamycin and/or amphotericin B
5. Use or expected use of antineoplastic drugs
6. No informed consent or unable to provide informed consent.
7. Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient's safety, or interfere with the interpretation of the study results.
8. Any illness which might affect patient's survival over the study follow-up period
9. History of skeletal muscle disease, either primary (i.e., myopathy) or secondary (i.e., ischemic) or any underlying myopathy such as myasthenia gravis, muscular dystrophy, etc.
10. Patients with active infectious disease and/or who are known to have tested positive for HIV, HTLV, HBV-sAg, HCV, CMV and/or syphilis
11. Cardiogenic shock or severe compromise in left ventricular systolic function defined as ejection fraction lower than 20 %.
12. History of intolerance to amiodarone.
13. End stage renal disease
14. Contraindication for MRI
15. Any significant laboratory abnormality which will in the investigator's opinion interfere with the patient's ability to comply with the protocol, compromise the patient's safety, or interfere with the interpretation of the study result.
16. Inability to identify the infarct area intra operatively

ARM - B

1. Previous angiogenic therapy or myocardial laser therapy
2. History of cancer within 5 years
3. Cardiogenic shock or severe compromise in left ventricular systolic function defined as ejection fraction lower than 20 %.
4. Left Ventricular Ejection Fraction ≥ 40%.
5. Known sensitivity to gentamycin and/or amphotericin B
6. Use or expected use of antineoplastic drugs
7. No informed consent or unable to provide informed consent
8. Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
9. Any illness which might affect patient's survival over the study follow-up period
10. History of skeletal muscle disease, either primary (i.e., myopathy) or secondary (i.e.,ischemic) or any underlying myopathy such as myasthenia gravis, muscular dystrophy, etc.
11. Patients with active infectious disease and/or who are known to have tested positive for HIV, HTLV, HBV-sAg, HCV, CMV and/or syphilis
12. Poor candidates for coronary artery bypass surgery
13. Patients who are in need of emergency bypass surgery
14. History of prior coronary artery bypass surgery
15. Patients with severe valvular heart disease
16. History of intolerance to amiodarone
17. End stage renal disease
18. Pregnancy
19. Contraindication for MRI
20. Any significant laboratory abnormality which will in the investigator's opinion interfere with the patient's ability to comply with the protocol, compromise the patient's safety, or interfere with the interpretation of the study result.
21. Inability to identify infarct area intra operatively.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel P. Lasala, M.D., Principal Investigator — TCA Cellular Therapy, LLC
Locations (1):
- TCA Cellular Therapy, LLC, Covington, Louisiana, United States